CLINICAL TRIAL: NCT00268541
Title: Physical Activity, Insulin Resistance and Adipose Tissue Gene Expression in the Offspring of Patients With Type 2 Diabetes
Brief Title: Physical Activity, Insulin Resistance and Function of Fat Tissue in the Offspring of Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 03BI004; BHF Project Grant PG/03/145
Record Dates: First submitted 2005-12-21; First posted 2005-12-22 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Diseases
Keywords: exercise; physical activity; insulin resistance; adipose tissue; gene expression
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Motor Activity; Insulin Resistance | interventions — Exercise

INTERVENTIONS:
Behavioral: Physical activity

SUMMARY:
Offspring of patients with type 2 diabetes have increased risk of developing diabetes and are typically more insulin resistant than their peers with no diabetes family history. We have recently demonstrated that, in contrast to their sedentary counterparts, physically active offspring are not insulin resistant. In the proposed controlled clinical study, we will examine the effects of a moderate exercise programme on insulin resistance, and other metabolic risk factors, in sedentary offspring and matched control subjects. We hypothesise that offspring will exhibit an augmented response to exercise, thereby normalising their predisposition to an adverse metabolic profile. We will also investigate expression of adipokines and other genes in adipose tissue to determine whether these contribute to the increased insulin resistance observed in offspring and whether they are influenced by exercise. The results will help to determine the efficacy of exercise in normalising metabolism in offspring and will help elucidate the mechanisms involved.

ELIGIBILITY:
Inclusion Criteria:

* 2 subject groups - 'control' and 'offspring'
* Offspring - at least 1 parent diagnosed with type 2 diabetes before age 65
* Controls - no history of type 2 diabetes in 1st or 2nd degree relatives
* In generally good health
* Non-smoker
* Fasting glucose < 7 mmol/l
* Blood pressure <160/90 mm Hg
* No established CHD (e.g. MI, stroke, CABG, PCTA)

Exclusion Criteria:

* Established CHD (e.g. MI, stroke, CABG, PCTA)
* diabetes
* smoking
* hypertension (BP > 160/90 mmHg)
* pregnancy

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80
Dates: Start 2004-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Insulin resistance at 8 weeks
Risk markers for cardiovascular disease/diabetes at 8 weeks
Adipose tissue gene expression at 8 weeks

SECONDARY OUTCOMES:
Fitness at 8 weeks
Body composition/adiposity at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jason MR Gill, BSc MSc PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom

REFERENCES:
- [Background] Higgins S, Gill JM, Janilionyte R, Caslake MJ, Malkova D. Physical activity, dietary intake and metabolic risk factors in non-diabetic daughters of patients with type II diabetes. Prev Med. 2005 Feb;40(2):145-51. doi: 10.1016/j.ypmed.2004.05.004. PMID 15533523
- [Derived] Barwell ND, Malkova D, Moran CN, Cleland SJ, Packard CJ, Zammit VA, Gill JM. Exercise training has greater effects on insulin sensitivity in daughters of patients with type 2 diabetes than in women with no family history of diabetes. Diabetologia. 2008 Oct;51(10):1912-9. doi: 10.1007/s00125-008-1097-6. Epub 2008 Jul 29. PMID 18663427